CLINICAL TRIAL: NCT00086775
Title: Phase II Trial Comparing Combination Treatment With Fludarabine and Alemtuzumab to Fludarabine and Rituximab in Patients With B-Cell Chronic Lymphocytic Leukemia Requiring Treatment After First Line Therapy
Brief Title: Fludarabine Combined With Either Alemtuzumab or Rituximab in Treating Patients With Refractory or Relapsed B-Cell Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: BRLX-FLUCAM106; CDR0000365631 (Registry Identifier: PDQ (Physician Data Query)); BRLX-STA1-03-058; OHSU-HEM-03050-P; DMS-F0334
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2009-10

CONDITIONS: Leukemia
Keywords: refractory chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab; Rituximab; fludarabine phosphate

INTERVENTIONS:
Biological: alemtuzumab
Biological: rituximab
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine, work in different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies, such as alemtuzumab and rituximab, can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Combining chemotherapy with monoclonal antibody therapy may kill more cancer cells. It is not yet known whether fludarabine is more effective when combined with alemtuzumab or with rituximab in treating chronic lymphocytic leukemia.

PURPOSE: Randomized phase II trial to compare the effectiveness of combining fludarabine with either alemtuzumab or rituximab in treating patients who have refractory or relapsed B-cell chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the complete response rate in patients with refractory or relapsed B-cell chronic lymphocytic leukemia treated with fludarabine and alemtuzumab vs fludarabine and rituximab.

Secondary

* Compare the overall response rate in patients treated with these regimens.
* Compare 1-year survival of patients treated with these regimens.
* Compare time to progression in patients treated with these regimens.
* Compare duration of response in patients treated with these regimens.
* Compare the adverse event profile of these regimens in these patients.
* Compare the molecular response rate in patients treated with these regimens.
* Compare lymphocyte and lymphocyte subset recovery (CD3, CD3/CD4, CD3/CD8, CD20) in patients treated with these regimens.
* Compare the time to complete response in patients treated with these regimens.
* Compare the rate of cytomegalovirus reactivation and time to reactivation in patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to prior treatment with fludarabine (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive fludarabine IV over 30 minutes on days 1-5. At least 30 minutes before fludarabine administration, patients receive alemtuzumab subcutaneously (SC) on days 1-5.
* Arm II: Patients receive fludarabine as in arm I. At least 30 minutes before fludarabine administration, patients receive rituximab IV on days 1 and 4 of course 1 and on day 1 only in subsequent courses.

In both arms, treatment repeats every 28 days for 4-6 courses in the absence of disease progression or unacceptable toxicity. An interim assessment is performed during course 4. Patients achieving a partial response or stable disease receive 2 additional courses of therapy (for a total of 6 courses). Patients achieving a complete response (CR) do not receive further treatment beyond CR.

Patients are followed weekly for 2 months, monthly for 6 months, every 2 months for 6 months, and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 150 patients (75 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of B-cell chronic lymphocytic leukemia (CLL), defined as:

  * Peripheral lymphocyte count > 5,000/mm^3
  * Clonal CD5-, CD19-, and CD23-positive lymphocytes
* Refractory to OR relapsed after prior first-line therapy
* No CNS involvement with CLL

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative

Renal

* Creatinine ≤ 1.5 times ULN

Immunologic

* No active cytomegalovirus
* No prior fludarabine-associated autoimmune hemolytic anemia or immune thrombocytopenic purpura
* No active infection requiring treatment with antibiotic, antiviral, or antifungal agents
* No prior significant allergic reaction to antibody therapies that required therapy to be discontinued
* HIV negative

Other

* No active secondary malignancy
* No other concurrent severe diseases or mental disorders
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior alemtuzumab and/or rituximab
* No prior bone marrow transplantation
* No concurrent thrombopoietin or pegfilgrastim

Chemotherapy

* More than 3 weeks since prior fludarabine

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 3 months since prior investigational drugs
* No other concurrent cytotoxic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-07; Primary Completion 2005-06 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann S. LaCasce, MD, Study Chair — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Jackson Oncology Associates, PLLC, Jackson, Mississippi
  - Cancer Institute of New Jersey at Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania